CLINICAL TRIAL: NCT05292287
Title: Remote Maintenance Cardiac Rehabilitation: a Randomised Feasibility Study
Brief Title: Remote Maintenance Cardiac Rehabilitation
Acronym: MAINTAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coventry University (Other)
Responsible Party: Principal Investigator, Francesca Denton, Chief Investigator, Coventry University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 302243; 121990 (Other: Coventry University Ethics)
Record Dates: First submitted 2021-12-16; First posted 2022-03-23 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Coronary Heart Disease
Keywords: Coronary Heart Disease; Exercise Maintenance; Cardiac Rehabilitation; Home-based Exercise; Wearable Activity Monitor
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The researcher carrying out the follow up assessments will be blinded to the arm participants have been randomised to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based Watch Intervention (Experimental): The home-based watch group will receive an exercise consultation with an exercise physiologist followed by check-in sessions at 1-month, 3-months, 6-months, and 12-months post-randomisation to set and review exercise and physical activity goals. They will wear a Polar Ignite wearable activity monitor which will help to monitor and guide their exercise sessions. Text-message feedback will be provided by an exercise physiologist based on information gathered from exercise sessions recorded on the watch by the participant.
  Interventions: Device: Polar Ignite Wearable Activity Monitor
- Best Practice Usual Care Control (No Intervention): No intervention will be administered. Best practice usual care and activity.

INTERVENTIONS:
Device: Polar Ignite Wearable Activity Monitor — A wearable activity monitor capable of monitoring outcomes relating to physical activity sedentary time, heart rate, and sleep quality. The watch synchronises to a corresponding mobile app called Polar Flow- Sync and Analyze or to the Polar FlowSync data transfer software on a computer.
  Arms: Home-based Watch Intervention

SUMMARY:
The investigators would like to test the feasibility of a remotely prescribed and monitored exercise program in people with coronary heart disease, using a wearable activity device and text message support, compared to usual care after completing cardiac rehabilitation. One group will use a Polar Ignite watch to guide them through exercise sessions at home and will receive text message feedback. The other group will be asked to continue their routine as usual. Assessments of both groups will happen after the completion of cardiac rehabilitation and at three follow-up time points of three, six, and twelve months. The aim of these treatments is to see if the investigators can help people to maintain their exercise adherence and coronary heart disease risk factor management after completing cardiac rehabilitation.

DETAILED DESCRIPTION:
Following the completion of centre-based cardiac rehabilitation (CR), lifetime adoption of physical activity (PA) and adherence to exercise is often poor. Wearable activity monitors may be a tool to remotely prescribe and monitor PA and exercise to promote long term behaviour change. This research aims to assess the feasibility of conducting a randomised controlled trial (RCT) testing a remotely prescribed and monitored long-term maintenance exercise programme in cardiac rehabilitation graduates with coronary heart disease (CHD). 30 participants with CHD will be recruited to a 12-month feasibility RCT and randomised into 2 arms: 1) a home-based watch intervention group and 2) a best practice usual care control group. The intervention group will receive an initial exercise consultation, personalised exercise prescription delivered via a Polar Ignite watch, and monitoring via check-ins and feedback text-message support with a clinical exercise physiologist. The control group will receive no intervention. All participants will undergo assessment at baseline (following the completion of CR) and at 3 follow up time points including 3-, 6- and 12-months. The primary outcome will be to assess feasibility and other process-related outcomes. The secondary outcomes will include exercise capacity, physical activity and sedentary behaviour, exercise time, cardiovascular disease risk, quality of life, depression, anxiety, self-efficacy, patient activation, health utility, health and social care resource use, cost, and adverse and serious adverse events. Semi-structured interviews will be conducted at 3-, 6-, and 12-months post-randomisation to explore the views, perceptions, acceptability, and experiences of the remotely prescribed and monitored exercise intervention and trial procedures. Participants who drop out or choose not to participate will be offered a semi-structured interview or a questionnaire, respectively, to understand feasibility. Overall, there is a need to support people post-CR to remotely maintain PA and exercise behaviour for secondary prevention of CHD particularly during the era of government-enforced restrictions or lockdowns due to the COVID-19 pandemic. The MAINTAIN study will assess the feasibility of longer-term remote prescription and monitoring of maintenance exercise following CR using a wearable activity monitor and text message support compared to best practice usual care for people diagnosed with CHD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed coronary heart disease.
* Completed community cardiac rehabilitation.
* Clinically stable (symptoms and medication).
* Men and women aged over 18.
* Access to smartphone with Bluetooth capacity or a computer/laptop.
* Able to provide informed consent.

Exclusion Criteria:

* Absolute contraindications to exercise as per international clinical guidelines.
* Any serious mental health/cognitive issue that will prevent engagement with study procedures or increase the risk of exercise complications.
* Diagnosed atrial fibrillation or other arrhythmia preventing accurate heart rate measurement.
* Allergy to watch materials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Intervention feasibility assessed via recruitment rate. | Will be evaluated after the 12-month follow up assessment
  The investigators will complete enrolment logs to record the number of people who enrol in the study.
Intervention feasibility assessed via number of screened patients. | Will be evaluated after the 12-month follow up assessment
  The investigators will complete screening logs to record the number of eligible participants.
Intervention feasibility assessed via number of patients randomised. | Will be evaluated after the 12-month follow up assessment
  The investigators will complete randomisation logs to record the number of participants randomised to both groups.
Intervention feasibility assessed via number of patients retained in the study. | Will be evaluated after the 12-month follow up assessment
  The investigators will assess the number of participants who withdraw or stay within the study.
Adherence to the prescribed exercise sessions. | Will be evaluated after the 12-month follow up assessment.
  The investigators will collect exercise session data recorded by the Polar Ignite watches worn by the participants in the intervention arm. The percentage of prescribed exercise sessions completed will be assessed.
Adherence to the prescribed exercise sessions' intensity. | Will be evaluated after the 12-month follow up assessment.
  The investigators will collect exercise session data recorded by the Polar Ignite watches worn by the participants in the intervention arm. The percentage of exercise time completed at the correct intensity will be assessed.
Adherence to the prescribed exercise sessions' duration. | Will be evaluated after the 12-month follow up assessment.
  The investigators will collect exercise session data recorded by the Polar Ignite watches worn by the participants in the intervention arm. The percentage of exercise time completed at the correct duration will be assessed.
Trial acceptability of the interventions and trial procedures via participant interviews | Interviews at 3 months
  Qualitative semi-structured interviews carried out with control and intervention participants as well as interviews with participants who withdraw from the study.
Trial acceptability of the interventions and trial procedures via participant interviews | Interviews at 6 months
  Qualitative semi-structured interviews carried out with control and intervention participants as well as interviews with participants who withdraw from the study.
Trial acceptability of the interventions and trial procedures via participant interviews | Interviews at 12 months
  Qualitative semi-structured interviews carried out with control and intervention participants as well as interviews with participants who withdraw from the study.

SECONDARY OUTCOMES:
Exercise capacity determined using an Incremental Shuttle Walk Test (ISWT). | Baseline, 3-, 6- and 12 month follow up post randomisation
  To assess heart rate and rating of perceived exertion over a 15 meter shuttle walk. Increases in distance walked indicates a higher exercise capacity. Changes in distance walked will be compared to participants randomised to the intervention vs the control group over time.
Physical activity and sedentary behaviour | The Actigraph will be worn during the baseline assessment and the 3-, 6, and 12-month follow up post randomisation.
  Using an Actigraph to measure free-living sedentary behaviour and physical activity behaviour. Changes in physical activity and sedentary behaviour will be compared to participants randomised to the intervention vs the control group over time.
Exercise frequency and intensity | It will be completed monthly from baseline to the 12-month follow up period to assess change over time.
  The Godin Leisure Time Exercise Questionnaire will be completed monthly to assess the frequency of 3 different exercise intensities over a week. Changes in exercise frequency and intensity will be compared to participants randomised to the intervention vs the control group over time. The questionnaire is broken down into strenuous, moderate, and mild physical activity completed in bouts of 15 minutes or more over the last week. A higher score indicates a more active individual and a lower score indicates a less active individual.
Cardiovascular disease risk using the Second Manifestations of Arterial disease (SMART) risk score | Measured at baseline, 3-, 6- and 12-month follow up
  A score taking into account cardiovascular history, smoking, blood pressure, and measures from blood samples including a full lipid profile, estimated glomerular filtration rate and high-sensitivity C-reactive protein. It identifies patients at a high risk of a reoccurring vascular event within 10 years. Changes in the risk score will be compared to participants randomised to the intervention vs the control group over time.
Cardiac specific quality of life using the MacNew Quality of Life Questionnaire | Baseline, 3-, 6-, and 12-months post randomisation.
  Using the MacNew Quality of Life Questionnaire to assess health-related quality of life. 1 indicates low health-related quality of life and 7 indicates high quality of life. Scores will be compared between participants randomised to the intervention vs the control group over time.
Depression using the Patient Health Questionnaire (PHQ-9) | Baseline, 3-, 6-, and 12-months post randomisation.
  Scores represent mild (0-5, moderate (6-10), moderately severe (11-15) and severe depression (16-20). Scores will be compared between participants randomised to the intervention vs the control group over time.
Anxiety using the Generalised Anxiety Disorder 7-item Scale (GAD-7) | Baseline, 3-, 6-, and 12-months post randomisation.
  A self report questionnaire to measure generalised anxiety disorder. Scores represent mild (0-5), moderate (6-10), moderately severe anxiety (11-15), and severe anxiety (15-21). Scores will be compared between participants randomised to the intervention vs the control group over time.
Self efficacy using the General Self-Efficacy Scale (GSE) | Baseline, 3-, 6-, and 12-months post randomisation.
  A 10-item psychometric scale to assess optimistic self-beliefs to cope with a range of life demands. Total scores can range from 10 up to 40. A higher score indicates a higher level of self-efficacy. Scores will be compared between participants randomised to the intervention vs the control group over time.
Patient activation using the Patient Activation Measure | Baseline, 3-, 6-, and 12-months post randomisation.
  Higher levels of activation are linked to positive health behaviours and outcomes. Scores will be compared between participants randomised to the intervention vs the control group over time.
Health utility using the EQ-5D-5L | Baseline, 3-, 6-, and 12-months post randomisation.
  The responses to the questionnaire can be converted into a health utility score using 5 levels to define a health state. Scores will be compared between participants randomised to the intervention vs the control group over time.
Health and social care resource use using the Client Service Receipt Inventory (CSRI) | Baseline, 3-, 6-, and 12-months post randomisation.
  We will use a health and social care resource use questionnaire to examine the feasibility of collecting these data and refine resource use schedules for use in a definitive trial. We will also test the feasibility of collecting patient-reported health outcome data. Scores will be compared between participants randomised to the intervention vs the control group over time.
Cost of the study | Baseline, 3-, 6-, and 12-months post randomisation.
  Cost of staff, the facility, consumables etc. of delivering active and control interventions. Costs will be compared between participants randomised to the intervention vs the control group.
Safety assessed via adverse and serious adverse events | Baseline, 3-, 6-, and 12-months post randomisation.
  Events will be documented in accordance with Good Clinical Practice (GCP). Adverse and serious adverse events will be compared between participants randomised to the intervention vs the control group over time.

CONTACTS AND LOCATIONS:
Overall Officials: Gordon McGregor, PhD, Principal Investigator — Coventry University
Locations (1):
- Atrium Health Limited, Coventry, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Denton F, Waddell A, Kite C, Hesketh K, Atkinson L, Cocks M, Jones H, Randeva H, Davenport N, Powell R, Clark C, Kyrou I, Harwood AE, McGregor G. Remote maintenance cardiac rehabilitation (MAINTAIN): A protocol for a randomised feasibility study. Digit Health. 2023 Feb 15;9:20552076231152176. doi: 10.1177/20552076231152176. eCollection 2023 Jan-Dec. PMID 36818155